CLINICAL TRIAL: NCT04264338
Title: The Validity of the Thyromental Height Test as a Predictor of the Difficult Airway: A Prospective Comparative Study With Interincisor Distance, Thyromental Distance, Sternomental Distance & Modified Mallampati Test
Brief Title: Thyromental Height Test as a Predictor of Difficult Airway:
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU & pain management. Kasralainy Faculty of medicine, Cairo University
Other Study IDs: MD-246-2019
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thyromental height test — Assessment of difficult airway

SUMMARY:
Anesthesia is increasingly safe. Major complications of airway management are no more common but still the most life-threatening condition amongst anesthesia practice and even medicine. Thyromental height test (TMHT) is an objective measure of the height between the anterior borders of the mentum and thyroid cartilage, measured while the patient is lying supine with the mouth closed. This study was designed to assess the validity of the TMHT as a single objective predictor for difficult laryngoscopy and to be compared to other objective measures.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I & II
* Scheduled for elective surgical procedures under general anesthesia using endotracheal with conventional laryngoscopy

Exclusion Criteria:

* Patients with a body mass index >35 kg/m2.
* Patients with neuromuscular disorders, craniofacial abnormalities, and abnormal dentition.
* Patients with airway diseases e.g cancer larynx or tongue, uncooperative patients, those who will need awake intubation and patients who will undergo emergency operations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients, aged from 18-60 years old, with ASA physical status I & II who will undergo elective surgical procedures under general anesthesia using endotracheal intubation using conventional laryngoscopy.
Sampling Method: Probability Sample
Enrollment: 612 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2020-08-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
validity of the TMHT in prediction of difficult airway in patients undergoing general anesthesia for elective surgeries using area under ROC curve for the TMHT. | baseline (before induction of general anesthesia)
Validity of TMHT in comparison with that of Modified Mallampati test (MMT) in prediction of difficult airway by comparing area under ROC curve for both tests. | baseline (before induction of general anesthesia)

IPD SHARING:
Plan to Share IPD: No